CLINICAL TRIAL: NCT07122882
Title: Integrated Genomics in Oncogene-driven Non-small Cell Lung Cancer With Acquired Resistance to Tyrosine Kinase Inhibitors
Brief Title: Integrated Genomics in Oncogene-driven NSCLC With Acquired Resistance
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chen-Yang Huang, Principal Investigator, M.D., Ph.D., Chang Gung Memorial Hospital
Other Study IDs: 202500569B0
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Oncogene-addicted Non Small Cell Lung Cancer; EGFR Mutation; ALK Fusion-positive Solid or CNS Tumors; ROS1 Fusion Positive; RET Fusion Positive; ERBB2 Mutation-Related Tumors; NTRK1 Fusion Positive; NTRK2 Fusion Positive; NTRK3 Fusion Positive; NRG1 Fusion; BRAF V600 Mutation; KRAS G12C Mutation; MET Exon 14 Skipping Mutation
Keywords: oncogene-driven NSCLC; acquired resistance; integrated genomics
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Solid tumor tissue sample, peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Oncogene-driven NSCLC with acquired resistance to tyrosine kinase inhibitor

SUMMARY:
Currently, tyrosine kinase inhibitor (TKI) remains the standard of care for oncogene-driven non-small cell lung cancer (NSCLC). However, almost all oncogene-driven NSCLCs would develop acquired resistance against TKI in clinical practice. Therefore, understanding the molecular mechanisms underlying the acquired resistance is a critical issue in lung cancer. Based on the literature, acquired resistance mechanism against EGFR TKI includes EGFR secondary mutation (T790M, C797X, L792X, G796X, L718Q, and exon 20 insertions), MET amplification, HER2 amplification, acquired gene fusions, and other complex alterations.

From the perspective of mutagenesis, the acquired resistance against TKI may be associated with APOBEC mutational processes, kataegis, chromothripsis, extrachromosomal DNA (ecDNA), and the interaction among them. However, still 30% to 50% of oncogene-driven NSCLCs had no identified mechanism attributed to the acquired resistance. Previous studies mostly used targeted-gene sequencing, which may overlook some structural variation and the transcriptomic dynamics. This study aims to investigate the genomic alterations, mutational processes, and the transcriptomic landscape underlying the acquired resistance using integrated genomics.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC, with at least one of the known oncogene mutation prior to systemic treatment: EGFR exon 18-21 activating mutation, MET exon-14-skipping mutation, ERBB2 activating mutation, ALK fusion, ROS1 fusion, RET fusion, NTRK1 fusion, NTRK2 fusion, NTRK3 fusion, BRAF V600 mutation, or KRAS G12C mutation
2. Patient had received tyrosine kinase inhibitor (TKI) with progressive disease, as assessed by the treating physician
3. Had tumor tissue available for DNA extraction and sequencing.
4. Eligible for withdrawal of a blood sample for DNA extraction and sequencing.

Exclusion Criteria:

1. Patient had not received TKI or did not have documented disease progression during TKI treatment.
2. Tumor tissue was unavailable for DNA extraction or the DNA quality did not meet the sequencing requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have histologically confirmed NSCLC, with at least one of the known oncogene mutation at baseline (EGFR exon 18-21 activating mutation, MET exon-14-skipping mutation, ERBB2 activating mutation, ALK fusion, ROS1 fusion, RET fusion, NTRK1 fusion, NTRK2 fusion, NTRK3 fusion, BRAF V600 mutation, or KRAS G12C mutation), and have documented disease progression during TKI treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-11 (Estimated); Study Completion 2028-05-11 (Estimated)

PRIMARY OUTCOMES:
Genomic alterations associated with resistance to TKI | Through study completion, an average of 2 years
  Tissue-based whole-genome and transcriptomic analysis of oncogene-driven NSCLC with acquired resistance to TKI

IPD SHARING:
Plan to Share IPD: Undecided